CLINICAL TRIAL: NCT06419205
Title: A Phase 2 Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Clinical Activity of ADX-097 Administered Subcutaneously in Male and Female Participants Aged 18 Years or Older With IgAN, LN, or C3G
Brief Title: A Phase 2 Study to Evaluate the Safety, PD, PK, and Clinical Activity of ADX-097 in Participants With IgAN, LN or C3G
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: study closed prior to enrolling any patients.
Sponsor: Q32 Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADX-097-201
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-12

CONDITIONS: IgA Nephropathy; Lupus Nephritis (LN); C3 (Complement Component 3) Glomerulopathy
MeSH Terms: conditions — Glomerulonephritis, IGA; Lupus Nephritis; Complement Component 3 Deficiency, Autosomal Recessive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Other): Subcutaneous Infusions
  Interventions: Drug: ADX-097

INTERVENTIONS:
Drug: ADX-097 — Open Label

SUMMARY:
A Phase 2 Study to Evaluate the Safety, Pharmacodynamics, Pharmacokinetics, and Clinical Activity of ADX-097 Administered Subcutaneously in Male and Female Participants Aged 18 Years or Older With Immunoglobulin A Nephropathy (IgAN), Lupus Nephritis (LN), or Complement Component 3 Glomerulopathy (C3G)

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants aged ≥18 years.
2. Urine protein ≥ 0.75 g/24 hours or uPCR ≥ 0.5g/g
3. Screening eGFR ≥30 mL/min/1.73m2 calculated by the Chronic Kidney Disease Epidemiology Collaboration creatinine equation (CKD-EPI GFR).
4. Participants receiving a RAAS inhibitor must have been on a stable dose (at the maximum recommended dose according to local guidelines or maximum tolerated dose) for at least 12 weeks prior to Study Day 1 that is projected to remain stable during the study.
5. Participants receiving a sodium-glucose cotransporter-2 (SGLT2) inhibitor or sparsentan must have been on a stable dose for at least 12 weeks prior to Study Day 1 that is projected to remain stable during the study.
6. Kidney biopsy-proven diagnosis of IgAN within 52 week; LN within 12 weeks or C3G within 52 weeks of Day 1 and with evidence of C3 fragment deposition.

Key Exclusion Criteria

1. A ≥50% decline in eGFR within 3 months before screening.
2. Concomitant significant renal disease other than IgAN, C3G, or LN.
3. Uncontrolled hypertension, defined as systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥90 mmHg, despite antihypertensive treatment.
4. Kidney, other solid organs, or bone marrow transplantation prior to or expected to occur during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) to evaluate the safety of ADX-097 | 42 weeks
  Incidence of adverse events (AEs) to evaluate the safety of ADX-097 when administered to participants with IgAN, LN, or C3G

SECONDARY OUTCOMES:
Change from baseline in urine protein-to-creatinine ratio (uPCR) | 26 weeks
  To evaluate clinical activity of ADX-097 in participants with IgAN, LN, or C3G
Change from baseline in estimated glomerular filtration rate (eGFR) | 26 weeks
  To evaluate clinical activity of ADX-097 in participants with IgAN, LN, or C3G

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Denver, Denver, Colorado
  - Minneapolis, Minneapolis, Minnesota
  - Las Vegas, Las Vegas, Nevada
  - New York, New York, New York
  - Columbus, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No